CLINICAL TRIAL: NCT00305370
Title: Aripiprazole Associated With Methylphenidate in Children and Adolescents With Bipolar Disorder and ADHD: A Randomized Cross-Over Placebo Controlled Trial
Brief Title: Aripiprazole Associated With Methylphenidate in Children and Adolescents With Bipolar Disorder and ADHD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GPPG03-325b
Record Dates: First submitted 2006-03-19; First posted 2006-03-21 (Estimated); Last update posted 2008-08-07 (Estimated); Status verified 2006-03

CONDITIONS: Bipolar Disorder; Attention Deficit Hyperactivity Disorder
Keywords: clinical trial; aripiprazole; methylphenidate; Bipolar Disorder; Attention-Deficit Hyperactivity Disorder; ADHD
MeSH Terms: conditions — Bipolar Disorder; Attention Deficit Disorder with Hyperactivity | interventions — Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole

SUMMARY:
There is a scarcity of clinical trials assessing the effects of medications in children with bipolar disorder. This study aims to assess the efficacy of Aripiprazole associated with Methylphenidate (MPH)for the treatment of children and adolescents with bipolar disorder comorbid with ADHD who improve in maniac symptoms while receiving aripiprazole but did not have an adequate response in ADHD symptoms. The study design is a 4-week randomized, double blind, cross-over group trial. Patients were randomized to aripiprazole + MPH or aripiprazole + placebo. The main hypothesis is: Aripiprazole + MPH will significantly reduce ADHD scores compared to aripiprazole + placebo.

DETAILED DESCRIPTION:
Bipolar disorder (BD) is a chronic disorder that severely affects the normal development of children and adolescents. The disorder is associated with high rates of suicide and high-risk behaviors like sexual promiscuity and drug abuse. Bipolar disorder in children is also associated with high rates of comorbidity, especially with Attention-Deficit Hyperactivity Disorder (ADHD). There is a scarcity of clinical trials assessing the effects of medications in children with BD. Moreover, the frequent presence of comorbid ADHD might determine lower response to treatment. Aripiprazole is a novel anti-psychotic drug. Its mechanism of action seems to be related to a stabilization of dopaminergic transmission, acting as a partial agonist especially in dopaminergic D2 receptors. It also has effects in 5-HT1a serotonergic receptors. Thus, it might have a promising effect in children and adolescents with comorbid BD and ADHD. A retrospective chart review, recently published, suggests the efficacy of this drug in children with BD. This study aims to assess the efficacy of Aripiprazole associated with Methylphenidate (MPH) for the treatment of 20 children and adolescents (age range: 8 to 17 years-old) with Bipolar Disorder comorbid with ADHD who improve in maniac symptoms while receiving aripiprazole but did not have an adequate response in ADHD symptoms. The study design is a 4-week randomized, double blind, cross-over group trial. Patients were randomized to aripiprazole + MPH or aripiprazole + placebo. The hypotheses are: 1) Aripiprazole + MPH will significantly reduce ADHD scores compared to aripiprazole + placebo. 2) Patients receiving aripiprazole + MPH will not deteriorate in maniac symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age: 8 -17
* BD type I or II comorbid with ADHD
* Reduction of maniac symptoms (30% reduction in the YMRS scores and/or CGI scores ≤ 2)while using aripiprazole during a previous study (NCT00116259)without improvement of ADHD symptoms (reduction in ADHD symptoms < 30% in the SNAP-IV). Those receiving placebo in the previous protocol will receive a 6- week open label treatment with aripiprazole. The same threshold for reducing maniac symptoms and absence of response in ADHD symptoms will be used.

Exclusion Criteria:

* IQ < 70
* Pregnancy or absence of a contraceptive method in fertile girls
* Diagnoses: pervasive development disorder, schizophrenia, drug abuse or dependency
* Risk of suicide or homicide
* Clinical condition that might interfere in the study
* Known sensibility to aripiprazole

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2005-08; Primary Completion 2008-01 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Scores in the SNAP-IV (ADHD)
Scores in the Young Mania Rating Scale (BD)
Weight

SECONDARY OUTCOMES:
Scores in CGI
Scores in the CMRS-P
Scores in the CDRS
Scores in the Kutcher Adolescent Depression Scale
Scores of quality of life (YQOL-R)
Report of side events

CONTACTS AND LOCATIONS:
Overall Officials: Luis A Rohde, MD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- ADHD Outpatient Program, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Scheffer RE, Kowatch RA, Carmody T, Rush AJ. Randomized, placebo-controlled trial of mixed amphetamine salts for symptoms of comorbid ADHD in pediatric bipolar disorder after mood stabilization with divalproex sodium. Am J Psychiatry. 2005 Jan;162(1):58-64. doi: 10.1176/appi.ajp.162.1.58. PMID 15625202
- [Result] Biederman J, McDonnell MA, Wozniak J, Spencer T, Aleardi M, Falzone R, Mick E. Aripiprazole in the treatment of pediatric bipolar disorder: a systematic chart review. CNS Spectr. 2005 Feb;10(2):141-8. doi: 10.1017/s1092852900019489. PMID 15685125
- [Derived] Zeni CP, Tramontina S, Ketzer CR, Pheula GF, Rohde LA. Methylphenidate combined with aripiprazole in children and adolescents with bipolar disorder and attention-deficit/hyperactivity disorder: a randomized crossover trial. J Child Adolesc Psychopharmacol. 2009 Oct;19(5):553-61. doi: 10.1089/cap.2009.0037. PMID 19877980